CLINICAL TRIAL: NCT01065519
Title: Assessment of Vessel Healing After DES Implantation With STEMI, NSTEMI and Stable/Unstable Angina Patients: a Randomized Study Between Everolimus and Biolimus A9-eluting Stents: an Optical Coherence Tomography (OCT) and Intravascular Ultrasound Tissue Characterisation (IVUS-TC) Study
Brief Title: STACCATO: Stent sTrut Apposition and Coverage in Coronary ArTeries: an Optical Coherence Tomography (OCT) Study
Acronym: STACCATO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2009-010923-14
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2009-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary stent; Optical coherence tomography; Intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): drug-eluting stent
  Interventions: Device: Xience V everolimus eluting stent
- 2 (Active Comparator): Biolimus A9-eluting Biomatrix stent
  Interventions: Device: Biolimus A9-eluting Biomatrix stent

INTERVENTIONS:
Device: Xience V everolimus eluting stent — Xience V everolimus eluting stent
  Arms: 1
Device: Biolimus A9-eluting Biomatrix stent — Biolimus A9-eluting Biomatrix stent
  Arms: 2

SUMMARY:
Assessment of vessel healing after DES implantation in STEMI, NSTEMI and stable/unstable angina patients: a randomized comparison between everolimus and biolimus A9-eluting stents: an optical coherence tomography (OCT) and intravascular ultrasound-tissue characterisation (IVUS-TC) study.

Plaque characterisation substudy: Assessment of culprit lesions in different subsets of patients (STEMI, NSTEMI and stable/unstable angina) by use of optical coherence tomography (OCT) and intravascular ultrasound tissue characterisation (IVUS-TC).

DETAILED DESCRIPTION:
1. The use of DES in STEMI and NSTEMI is still a matter of intense debate. Reassuring data of trials, meta-analyses and registries conflict with reports of delayed arterial healing and higher risk of stent thrombosis after DES implantation in ACS patients. Heterogeneity in healing (bad healing at the site of the necrotic core), stent strut malapposition and plaque prolapse are all proposed as possible causes for a higher risk of stent thrombosis. Furthermore, next generation DES claims a better safety profile in comparison to first-generation DES.
2. Thus far, our information on tissue characterisation of coronary plaques prone to rupture, relies on histopathology data. Recently, new invasive coronary imaging techniques; radiofrequency intravascular ultrasound (RF-IVUS) and optical coherence tomography (OCT) provide new possibilities for in vivo assessment of coronary plaques.

Aims:

1. To evaluate vessel healing, expressed as stent strut coverage and stent strut apposition assessed with OCT at 9 months after PCI and compare between everolimus Xience V (Abbott Vascular, Santa Clara, CA) and biolimus A9-eluting Biomatrix (Biosensors, Newport Beach, CA) stents, in 3 different groups of patient subsets (STEMI, NSTEMI and patients with stable/unstable angina).
2. To make, by use of OCT and IVUS-TC, a detailed characterisation of coronary lesions before PCI and to study the possible link between specific lesion characteristics (e.g. thin cap fibroatheroma, large necrotic core, extensive calcification,…) and outcome (risk of distal embolisation and myonecrosis in the short term, risk of bad strut coverage or risk of restenosis or stent thrombosis on longer term). To compare the performance of both technologies (OCT and IVUS-TC) in a direct way.
3. To assess, by use of OCT and IVUS-TC, the stented segment just after the intervention (assessment of stent expansion, stent strut apposition, detection of edge dissection, intraluminal thrombus) and correlate with angiographic and clinical outcomes. Again, the performance of both technologies will be compared in a direct way.
4. To study the influence of drug-eluting stent implantation in a 3-5 cm long segment of the coronary artery just distal to the implanted stent by use of OCT at baseline and at 9 months after stent implantation.

Methods: Patients undergoing PCI are recruited from 3 groups of patients: patients with STEMI (group I), patients with NSTEMI (group II) and patients with stable/unstable angina (group III). From each group, 20 patients are included. In each individual group, randomization between an everolimus-eluting stent and a biolimus A9-eluting stent is performed. All patients undergo IVUS-TC and OCT examination of the stented segment (and the 3 to 5 cm distal from the stented segment) just before and after stent implantation at the time of the index procedure. All patients undergo control angiography with OCT examination at 9 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. Written informed consent available
3. Patient eligible for percutaneous coronary intervention
4. patients with a single or multiple de novo lesion(s) from 3 different patient subsets (STEMI, NSTEMI, stable/unstable angina). Target reference vessel diameter measured by QCA: 2-4 mm

Exclusion Criteria:

1. Left ventricular ejection fraction of < 30%
2. Hemodynamic unstability (cardiogenic shock, life-threatening arrhythmias, inotropic support)
3. Impaired renal function (serum creatinine > 2.0 mg/dl)
4. Target lesion located in bifurcation
5. Lesion of the left main trunk > 50%, unprotected
6. Known allergies to antiplatelet, anticoagulation therapy, contrast media, everolimus or biolimus A9
7. Pregnant and/or breast-feeding females or females who intend to become pregnant (pregnancy test required)
8. Patients with a life expectancy of less than one year
9. Patient currently enrolled in other investigational device or drug trial
10. Patient not able or willing to adhere to follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2016-01-14 (Actual)

PRIMARY OUTCOMES:
Stent strut coverage and stent strut apposition, assessed with OCT | 9 months

SECONDARY OUTCOMES:
Lumen Loss (in-stent) at 9 months In-segment Late Lumen Loss at 9 months Cumulative MACE rate at 9 months Stent thrombosis at all follow-ups Target lesion revascularisation Device succes | 9 months, 12 months, yearly until 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium